CLINICAL TRIAL: NCT01260909
Title: Real-Time MV/kV Image Guided Radiation Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PROS0038; SU-12132010-7282 (Other: Stanford University); R21CA153587 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Real-time kV/MV Prostate Imaging
  Interventions: Device: Real-time kV/MV Prostate Imaging

INTERVENTIONS:
Device: Real-time kV/MV Prostate Imaging — The kV images will be acquired using onboard kV X-Ray imaging system existing in the clinical linear accelerator (LINAC).
  Other Names: Image-guided radiation therapy; External beam radiotherapy

SUMMARY:
In current radiation therapy, imaging (typically, cone beam CT imaging or two orthogonal X-ray projection imaging) is done for patient setup before radiation dose delivery. Dose delivery typically takes 2 to 5 minutes depending on the delivery technique used for treatment. A tumor target may change its position during the dose delivery process. The goal of this project is develop a real-time imaging strategy to monitor the tumor position during dose delivery and evaluate its potential clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be drawn from available patient population that will be treated using IMRT/VMAT. The Stanford population of IMRT/VMAT will be taken as roughly representative of prospective IMRT patients and will not be subdivided by any additional characteristics.

Exclusion Criteria:

* The study population will be drawn from available patient population that will be treated using IMRT/VMAT. The Stanford population of IMRT/VMAT will be taken as roughly representative of prospective IMRT patients and will not be subdivided by any additional characteristics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate cancer patients at Stanford University
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To verify improved tumor targeting accuracy using IMRT (intensity modulated radiation therapy) and VMAT (volumetric modulated radiation therapy) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xing, Principal Investigator — Stanford University